CLINICAL TRIAL: NCT02218879
Title: Restoring Glutathione Synthesis With Tecfidera: An in Vivo H-MRS Single-Arm Study at 7T in Patients With Relapsing-Remitting Multiple Sclerosis
Brief Title: Restoring Glutathione Synthesis With Tecfidera: An in Vivo H-MRS Single-Arm Study at 7T in Patients With RR MS
Status: Terminated | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1403013581
Record Dates: First submitted 2014-08-12; First posted 2014-08-18 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with relapsing MS
  Interventions: Drug: Tecfidera

INTERVENTIONS:
Drug: Tecfidera — Oral Tecfidera 240 mg bid

SUMMARY:
The primary objective is to directly estimate brain glutathione concentrations in vivo using H-MRS at 7T before and after initiation of Tecfidera in established multiple sclerosis (MS) patients considering switching therapy or being treatment-naive (first line).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patients
* 18-60 years of age
* Diagnosis of multiple sclerosis, in accordance with the revised McDonald criteria (2010)
* Patients naive to MS therapy or patients switching from an FDA-approved MS therapy, including IFN-B formulations, Cop-1, Teriflunomide, and Fingolimod to BG-12
* Expanded Disability Status Scale (EDSS) score 0 to 5.5 inclusive

Exclusion Criteria:

* Primary progressive multiple sclerosis patients
* Patients with previous exposure or known allergies to fumarates
* MS patients switching from natalizumab, cyclophosphamide, or mitoxantrone to BG-12
* Contraindications for MRI/MRS
* Known presence of other neurological disorders that may mimic multiple sclerosis
* Pregnancy or lactation
* Requirement for chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* History of or currently active primary or secondary immunodeficiency
* Active infection, or history of or known presence of recurrent or chronic infection (e.g. hepatitis B or C, HIV, syphilis, tuberculosis_
* History of progressive multifocal leukoencephalopathy
* Contraindications to or intolerance of oral or intravenous (IV) corticosteroids

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with a relapsing form of MS
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Glutathione Concentrations In Normal Appearing Gray Matter in Brain Measured by 7T Magnetic Resonance Imaging Scan | Before and 12 months after Tecfidera Initiation

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pelletier, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Juchem C, Swanberg KM, Prinsen H, Pelletier D. In vivo cortical glutathione response to oral fumarate therapy in relapsing-remitting multiple sclerosis: A single-arm open-label phase IV trial using 7-Tesla 1H MRS. Neuroimage Clin. 2023;39:103495. doi: 10.1016/j.nicl.2023.103495. Epub 2023 Aug 15. PMID 37651844